CLINICAL TRIAL: NCT01969838
Title: A Phase 3, Randomized, Double-blind Active-controlled Study Evaluating Momelotinib vs. Ruxolitinib in Subjects With Primary Myelofibrosis (PMF) or Post-Polycythemia Vera or Post-Essential Thrombocythemia Myelofibrosis (Post-PV/ET MF)
Brief Title: Momelotinib Versus Ruxolitinib in Subjects With Myelofibrosis
Acronym: Simplify 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-352-0101; 2013-002707-33 (EudraCT Number)
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Results first posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Primary Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide; ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Momelotinib (Experimental): Participants will receive momelotinib plus placebo to match ruxolitinib.
  Interventions: Drug: Momelotinib; Drug: Placebo to match ruxolitinib
- Ruxolitinib (Active Comparator): Participants will receive ruxolitinib plus placebo to match momelotinib.
  Interventions: Drug: Ruxolitinib; Drug: Placebo to match momelotinib

INTERVENTIONS:
Drug: Momelotinib — Momelotinib tablet administered orally once daily
  Other Names: GS-0387; CYT387
  Arms: Momelotinib
Drug: Ruxolitinib — Ruxolitinib tablets administered orally twice daily
  Arms: Ruxolitinib
Drug: Placebo to match momelotinib — Placebo to match momelotinib tablets administered orally once daily
  Arms: Ruxolitinib
Drug: Placebo to match ruxolitinib — Placebo to match ruxolitinib tablets administered orally twice daily
  Arms: Momelotinib

SUMMARY:
This study is to determine the efficacy of momelotinib (MMB) versus ruxolitinib (RUX) in participants with primary myelofibrosis (PMF) or post-polycythemia vera or post-essential thrombocythemia myelofibrosis (post-PV/ET MF) who have not yet received treatment with a Janus kinase inhibitor (JAK inhibitor).

Participants will be randomized to receive either MMB or ruxolitinib for 24 weeks during a double-blind treatment phase, after which they will be eligible to receive open-label MMB for up to an additional 216 weeks. After discontinuation of study medication, assessments will continue for 12 additional weeks, after which participants will be contacted for survival follow-up approximately every 6 months for up to 5 years from the date of enrollment or until study termination. For those participants planning to continue treatment with MMB following the end of the study, the Early Study Drug Discontinuation (ESDD), 30-day, 12-Week, and survival follow-up visits are not required.

ELIGIBILITY:
Key Inclusion Criteria:

* Palpable splenomegaly at least 5 cm below the left costal margin
* Confirmed diagnosis of PMF or post-PV/ET MF
* Requires myelofibrosis therapy, in the opinion of the investigator
* Classified as high risk OR intermediate-2 risk as defined by the International Prognostic Scoring System (IPSS) for PMF, or intermediate-1 risk (IPSS) associated with symptomatic splenomegaly, hepatomegaly, anemia (hemoglobin < 10.0 g/dL), and/or unresponsive to available therapy
* Acceptable laboratory assessment obtained within 14 days prior to the first dose of study drug:

  * Absolute neutrophil count (ANC) ≥ 0.75 x 10^9/L in the absence of growth factor in the prior 7 days
  * Platelet Count ≥ 50 x 10^9/L (≥ 100 x 10^9/L if aspartate aminotransferase [AST] or alanine aminotransferase [ALT] is ≥ 2 x the upper limit of the normal range [ULN]) in the absence of platelet transfusion(s) or thrombopoietin mimetics in the prior 7 days
  * Peripheral blood blast count < 10%
  * AST and ALT ≤ 3 x ULN (≤ 5 x ULN if liver is involved by extramedullary hematopoiesis as judged by the investigator or if related to iron chelator therapy that was started within the prior 60 days)
  * Calculated creatinine clearance (CrCL) of ≥ 45 mL/min
  * Direct bilirubin ≤ 2.0 x ULN
* Life expectancy of > 24 weeks
* Males and females of childbearing potential must agree to use protocol-specified method(s) of contraception
* Females who are nursing must agree to discontinue nursing before the first dose of study drug
* Able to understand and willing to sign the informed consent form

Key Exclusion Criteria:

* Prior splenectomy
* Splenic irradiation within 3 months prior to the first dose of study drug
* Eligible for allogeneic bone marrow or stem cell transplantation
* Uncontrolled inter-current illness, per protocol.
* Known positive status for human immunodeficiency virus (HIV)
* Chronic active or acute viral hepatitis A, B, or C infection, or a hepatitis B or C carrier
* Prior use of a JAK1 or JAK2 inhibitor
* Use of chemotherapy, immunomodulating therapy, biologic therapy, radiation therapy, or investigational therapy within 4 weeks of the first dose of study drug
* Presence of peripheral neuropathy ≥ Common Terminology Criteria for Adverse Events (CTCAE) Grade 2
* Unwilling or unable to undergo a magnetic resonance imaging (MRI) or computed tomography (CT) scan

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2013-12-06 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (114):
- United States (11):
  - Phoenix, Arizona
  - Escondido, California
  - Stanford, California
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - St Louis, Missouri
  - Durham, North Carolina
  - Seattle, Washington
- Australia (10):
  - Darlinghurst, New South Wales
  - Parkville, New South Wales
  - Saint Leonards, New South Wales
  - Brisbane, Queensland
  - Herston, Queensland
  - Adelaide, South Australia
  - Bedford Park, South Australia
  - Frankston, Victoria
  - Melbourne, Victoria
  - Perth, Western Australia
- Vienna, Vienna, Austria
- Belgium (4):
  - Charleroi, Hainaut
  - Antwerp
  - Leuven
  - Liège
- Bulgaria (5):
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Varna
- Canada (4):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Toronto, Ontario
- Czechia (3):
  - Hradec Králové, Vychodocesky KRAJ
  - Brno
  - Ostrava
- Denmark (2):
  - Aalborg
  - Herlev
- France (10):
  - Pierre-Bénite, Auvergne-Rhône-Alpes
  - Toulouse, Midi-pyrenees
  - Le Kremlin-Bicêtre
  - Lens
  - Lille
  - Marseille
  - Nantes
  - Paris
  - Pessac
  - Villejuif
- Germany (8):
  - München, Bavaria
  - Leipzig, Saxony
  - Dresden
  - Düsseldorf
  - Freiburg im Breisgau
  - Hamburg
  - Mainz
  - Mannheim
- Hungary (3):
  - Budapest
  - Debrecen
  - Kaposvár
- Israel (5):
  - Afula
  - Ashkelon
  - Haifa
  - Jerusalem
  - Tel Aviv
- Japan (9):
  - Ōgaki, Gifu
  - Kitaku Sapporo, Hokkaido
  - Osaka, Osaka
  - Ōsaka-sayama, Osaka
  - Bunkyo-ku, Tokyo
  - Fukushima
  - Kumamoto
  - Matsuyama
  - Okayama
- Netherlands (4):
  - Maastricht
  - Nijmegen
  - Rotterdam
  - Utrecht
- Poland (9):
  - Poznan, Greater Poland Voivodeship
  - Krakow, Lesser Poland Voivodeship
  - Lublin, Lublin Voivodeship
  - Warsaw, Mazowiekie
  - Gdansk, Pomeranian Voivodeship
  - Bialystok
  - Brzozów
  - Chorzów
  - Lodz, Łódź Voivodeship
- Romania (5):
  - Arad
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Iași
- Singapore, Singapore
- Seoul, South Korea
- Spain (6):
  - Majadahonda, Madrid
  - Pamplona, Navarre
  - Badalona
  - Barcelona
  - Valencia
  - Zaragoza
- Sweden (4):
  - Lund, Skåne County
  - Örebro
  - Stockholm
  - Uddevalla
- Kaohsiung City, Taiwan
- United Kingdom (8):
  - Leicester, England
  - London, England
  - Manchester, England
  - Newcastle upon Tyne, England
  - Oxford, England
  - Cardiff, Wales
  - Northern Ireland
  - Nottingham

REFERENCES:
- [Derived] Mesa RA, Talpaz M, Mazerolle F, Gorsh B, M'Hari M, Regnault A, Ellis C, Wang Z, Purser M, Liu T, Strouse B, Patnaik D. Time Without Transfusion Reliance (TWiTR): Integrating Survival Quality Into Myelofibrosis Treatment Strategies Based on the Phase 3 SIMPLIFY-1, SIMPLIFY-2, and MOMENTUM Trials. EJHaem. 2025 Jun 18;6(3):e70075. doi: 10.1002/jha2.70075. eCollection 2025 Jun. PMID 40535755
- [Derived] Harrison CN, Mesa R, Talpaz M, Gupta V, Gerds AT, Perkins A, Goh YT, Fox ML, McLornan D, Palmer J, Foltz L, Vannucchi A, Koschmieder S, Passamonti F, Lee SE, Ellis C, Strouse B, Gonzalez Carreras FJ, Oh ST. Longitudinal Assessment of Transfusion Intensity in Patients With JAK Inhibitor-Naive or -Experienced Myelofibrosis Treated With Momelotinib. Clin Lymphoma Myeloma Leuk. 2025 Mar;25(3):199-211. doi: 10.1016/j.clml.2024.10.001. Epub 2024 Oct 16. PMID 39516087
- [Derived] Verstovsek S, Mesa R, Gupta V, Lavie D, Dubruille V, Cambier N, Platzbecker U, Hus M, Xicoy B, Oh ST, Kiladjian JJ, Vannucchi AM, Gerds A, Egyed M, Mayer J, Sacha T, Kawashima J, Morris M, Huang M, Harrison C. Momelotinib long-term safety and survival in myelofibrosis: integrated analysis of phase 3 randomized controlled trials. Blood Adv. 2023 Jul 25;7(14):3582-3591. doi: 10.1182/bloodadvances.2022009311. PMID 37042865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 432 participants were randomized at 131 centers in 22 countries.
Pre-assignment Details: Participants were screened within 35 days after signing the informed consent form to determine eligibility for participation in the study. Participants who were not randomized within the 35 day screening window were screen failed. At randomization, participants were randomly assigned 1:1 to MMB plus RUX-placebo or RUX plus MMB-placebo.
Groups:
- Momelotinib (MMB): Participants received momelotinib plus placebo to match ruxolitinib.
  Momelotinib tablets were administered orally once daily at a starting dose of 200 mg. Additional available strengths included 100 mg and 150 mg.
  Placebo to match ruxolitinib tablets were administered orally twice daily.
- Ruxolitinib (RUX): Participants received ruxolitinib plus placebo to match momelotinib.
  Ruxolitinib tablets were administered orally twice daily (BID). The dose ranged from 5 to 20 mg BID and was dependent on platelet count, creatinine clearance, and transaminase levels.
  Placebo to match momelotinib tablets were administered orally once daily.
- MMB to MMB: After completion of the 24-week double-blind treatment phase, participants had the option to receive MMB in an open-label treatment phase for up to an additional 216 weeks. Participants randomized to the MMB group at study entry continued MMB in the open-label treatment phase at their current dose. Available MMB strengths were 100 mg, 150 mg and 200 mg.
- RUX to MMB: After completion of the 24-week double-blind treatment phase, participants had the option to receive MMB in an open-label treatment phase for up to an additional 216 weeks. Participants randomized to the RUX group who wished to remain in the study initiated MMB in the open-label treatment phase at the dose matching their equivalent MMB placebo dose. Available MMB strengths were 100 mg, 150 mg and 200 mg.
Period: Double-blind Phase
Arm/Group | Momelotinib (MMB) | Ruxolitinib (RUX) | MMB to MMB | RUX to MMB
Started | 215 (The MMB group is only applicable to the double-blind phase. Participants who complete the double-blind phase and continue to receive MMB in the open-label phase constitute the MMB to MMB group.) | 217 (The RUX group is only applicable to the double-blind phase. Participants who complete the double-blind phase and begin receiving MMB in the open-label phase constitute the RUX to MMB group.) | 0 (The MMB to MMB group is only applicable to the open-label phase.) | 0 (The RUX to MMB group is only applicable to the open-label phase.)
Completed | 188 | 208 | 0 | 0
Not Completed | 27 | 9 | 0 | 0
Not completed — Adverse Event | 10 | 4 | 0 | 0
Not completed — Death | 5 | 2 | 0 | 0
Not completed — Physician Decision | 5 | 1 | 0 | 0
Not completed — Subject Decision | 4 | 2 | 0 | 0
Not completed — Disease Progression | 2 | 0 | 0 | 0
Not completed — Symptomatic Spleen Growth | 1 | 0 | 0 | 0
Period: Open-label Phase
Arm/Group | Momelotinib (MMB) | Ruxolitinib (RUX) | MMB to MMB | RUX to MMB
Started | 0 (The MMB group is only applicable to the double-blind phase. Participants who complete the double-blind phase and continue to receive MMB in the open-label phase constitute the MMB to MMB group.) | 0 (The RUX group is only applicable to the double-blind phase. Participants who complete the double-blind phase and begin receiving MMB in the open-label phase constitute the RUX to MMB group.) | 171 (Of 188 participants in the MMB group who completed the double-blind phase, 171 entered the open-label phase to continue receiving MMB.) | 197 (Of 208 participants in the RUX group who completed the double-blind phase, 197 entered the open-label phase to begin receiving MMB.)
Completed (Defined as completing survival follow-up for a period of up to 5 years from randomization.) | 0 | 0 | 1 (The Sponsor terminated the study prior to subjects completing the 5 years of follow-up with the exception of a single subject. Subjects receiving MMB at the time of study termination were eligible to transition to an extended access study (SRA-MMB-4365) to continue MMB treatment.) | 0
Not Completed | 0 | 0 | 170 | 197
Not completed — Transferred to study SRA-MMB-4365 | 0 | 0 | 52 | 62
Not completed — Adverse Event | 0 | 0 | 37 | 49
Not completed — Disease Progression | 0 | 0 | 26 | 27
Not completed — Lack of Efficacy | 0 | 0 | 17 | 19
Not completed — Subject Decision | 0 | 0 | 14 | 15
Not completed — Death | 0 | 0 | 13 | 11
Not completed — Physician Decision | 0 | 0 | 9 | 14
Not completed — Non-compliance with Study Drug | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Momelotinib (MMB): Participants received momelotinib plus placebo to match ruxolitinib.
  Momelotinib: Momelotinib tablets were administered orally once daily at a starting dose of 200 mg. Additional available strengths included 100 mg and 150 mg.
  Placebo to match ruxolitinib: Placebo to match ruxolitinib tablets were administered orally twice daily.
- Ruxolitinib (RUX): Participants received ruxolitinib plus placebo to match momelotinib.
  Ruxolitinib: Ruxolitinib tablets were administered orally twice daily. The dose ranged from 5 to 20 mg BID and was dependent on platelet count, creatinine clearance, and transaminase levels.
  Placebo to match momelotinib: Placebo to match momelotinib tablets were administered orally once daily
- Total: Total of all reporting groups
Arm/Group | Momelotinib (MMB) | Ruxolitinib (RUX) | Total
Number analyzed (Participants) | 215 | 217 | 432
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 90 | 95 | 185
  >=65 years | 125 | 122 | 247
Age, Continuous [Median (Full Range); unit: years] | 67 [28 to 85] | 66 [25 to 86] | 66 [25 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 97 | 188
  Male | 124 | 120 | 244
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 191 | 194 | 385
  Unknown or Not Reported | 18 | 19 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 179 | 178 | 357
  Black or African American | 2 | 2 | 4
  Asian | 17 | 20 | 37
  Not Permitted | 15 | 16 | 31
  Other | 2 | 1 | 3
Transfusion Dependent [Count of Participants; unit: Participants]
  Yes | 53 | 52 | 105
  No | 162 | 165 | 327
Platelet Count (10^9/L) [Count of Participants; unit: Participants]
  < 100 | 18 | 23 | 41
  >= 100 and <= 200 | 66 | 63 | 129
  > 200 | 131 | 131 | 262
Weight [Median (Inter-Quartile Range); unit: kg] | 69.3 [62.9 to 80.0] | 71.4 [62.5 to 83.4] | 70.0 [62.8 to 82.0]
Height [Median (Inter-Quartile Range); unit: cm] | 170.0 [163.0 to 176.0] | 170.0 [162.0 to 177.0] | 170.0 [162.5 to 176.0]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 24.6 [22.0 to 26.7] | 24.9 [22.3 to 27.5] | 24.6 [22.2 to 27.2]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 10.5 [9.1 to 12.0] | 10.3 [9.2 to 11.9] | 10.4 [9.1 to 12.0]

OUTCOME MEASURES:

1. Primary Outcome: Splenic Response Rate at Week 24
Description: Splenic response rate at Week 24 is defined as the percentage of participants who achieved a spleen volume reduction of ≥ 35% from baseline at the Week 24 assessment as measured by MRI or CT.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Groups:
- Ruxolitinib (RUX): Participants received ruxolitinib plus placebo to match momelotinib.
  Ruxolitinib tablets were administered orally twice daily. The dose ranged from 5 to 20 mg BID and was dependent on platelet count, creatinine clearance, and transaminase levels.
  Placebo to match momelotinib tablets were administered orally once daily.
Arm/Group | Momelotinib (MMB) | Ruxolitinib (RUX)
Number analyzed (Participants) | 215 | 217
Participants
  Responder | 57 | 64
  Nonresponder | 158 | 153
Statistical Analysis 1: Comparison: Momelotinib (MMB) vs Ruxolitinib (RUX); Test type: Non-Inferiority — To evaluate the noninferiority of MMB over RUX, a conventional 2-sided confidence interval (CI) was calculated for the difference in splenic response rate (SRR) at Week 24: delta = prob(MMB) - 0.6*prob(RUX). If the lower bound of the 2-sided 95% CI for delta was greater than 0, MMB was declared noninferior to RUX in SRR at Week 24. The 2-sided 95% CI of delta was calculated based on stratum-adjusted Cochran-Mantel-Haenszel (CMH) proportions. This is the noninferiority proportion difference; p = 0.014, Cochran-Mantel-Haenszel; Proportion Difference - Stratified CMH = 0.09, 95% CI 2-sided [0.02 to 0.16]

2. Secondary Outcome: Total Symptom Score (TSS) Response Rate at Week 24
Description: Total symptom score (TSS) is defined as the percentage of participants who achieved a ≥50% reduction in TSS at Week 24 versus baseline as measured by the modified Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) v2.0 diary. Response rate was calculated using the average of the daily TSS from a consecutive 28-day period prior to Week 24, which had ≥20 daily TSS available.
  The modified MPN-SAF patient-reported outcome instrument consisted of 8 items assessing worst daily incidence of tiredness, filling up quickly, abdominal discomfort, night sweats, itching, bone pain, pain under ribs on left side, and inactivity. Scoring of the Total Symptom Score (TSS), in this study was based on 7 of these items, (range of 0-70,), excluding inactivity. These items assess the impact experienced by the participant in the 24 hours prior to completing the questionnaire. All items are measured using a 0 to 10 Numeric Rating Scale, with 0 corresponding to "Absent" and 10 being the worse
Time Frame: Week 24
Population: TSS rate analysis at Week 24 only included participants with TSS > 0 at baseline or with TSS = 0 at baseline but with TSS > 0 or missing at Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Momelotinib (MMB) | Ruxolitinib (RUX)
Number analyzed (Participants) | 211 | 211
Participants
  Responder | 60 | 89
  Nonresponder | 151 | 122
Statistical Analysis 1: Comparison: Momelotinib (MMB) vs Ruxolitinib (RUX); Test type: Non-Inferiority — To evaluate the noninferiority of MMB over RUX, a conventional 2-sided CI was calculated for the difference in TSS response rate at Week 24: delta = prob(MMB) - 0.67*prob(RUX). If the lower bound of the 2-sided 95% CI for delta was greater than 0, MMB was declared to be noninferior to RUX in TSS response rate at Week 24. The 2-sided 95% CI of delta was calculated based on stratum-adjusted Cochran-Mantel-Haenszel (CMH) proportions. This is called the noninferiority proportion difference; p = 0.98, Cochran-Mantel-Haenszel; Proportion Difference - Stratified CMH = 0.00, 95% CI 2-sided [-0.08 to 0.08]

3. Secondary Outcome: Rate of Red Blood Cell (RBC) Transfusions in the Double-blind Phase, (the Average Number of RBC Units Transfused Per Month Not Associated With Overt Bleeding)
Description: Rate of RBC transfusion was defined as the average number of RBC units transfused not associated with clinically overt bleeding per subject-month during the double-blind phase.
Time Frame: Baseline to Week 24
Measure: Median (Inter-Quartile Range); unit: units/month
Arm/Group | Momelotinib (MMB) | Ruxolitinib (RUX)
Number analyzed (Participants) | 215 | 217
units/month | 0.0 [0.0 to 0.2] | 0.4 [0.0 to 1.5]
Statistical Analysis 1: Comparison: Momelotinib (MMB) vs Ruxolitinib (RUX); Test type: Superiority; p < 0.001, Negative Binomial Model, Adjusted; Rate ratio = 0.28, 95% CI 2-sided [0.19 to 0.43] — A smaller ratio represents larger benefit

4. Secondary Outcome: RBC Transfusion Independence Rate at Week 24, (Defined as Absence of RBC Transfusions and no Hemoglobin Level Below 8 g/dL in the 12 Weeks Prior to Week 24, Excluding Cases Associated With Clinically Overt Bleeding)
Description: RBC transfusion independence is the percentage of participants who are transfusion independent at Week 24, defined as absence of RBC transfusions and no hemoglobin level below 8 g/dL in the 12 weeks prior to Week 24, excluding cases associated with clinically overt bleeding.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Momelotinib (MMB) | Ruxolitinib (RUX)
Number analyzed (Participants) | 215 | 217
Participants
  Responder | 143 | 107
  Nonresponder | 72 | 110
Statistical Analysis 1: Comparison: Momelotinib (MMB) vs Ruxolitinib (RUX); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Proportion Difference - Stratified CMH = 0.18, 95% CI 2-sided [0.09 to 0.26] — A larger proportion represents larger benefit

5. Secondary Outcome: RBC Transfusion Dependence Rate at Week 24. (Defined as Having Had at Least 4 Units of RBC Transfusions, or a Hemoglobin Level Below 8 g/dL in 8 Weeks Prior to Week 24 (Excluding Cases Associated With Clinically Overt Bleeding)).
Description: RBC transfusion dependence is the percentage of participants who are transfusion dependent at Week 24, defined as having had at least 4 units of RBC transfusions, or a hemoglobin level below 8 g/dL in 8 weeks prior to Week 24 (excluding cases associated with clinically overt bleeding). Participants with the last double-blind phase participation date prior to Day 162 (ie. missing at Week 24) were considered transfusion dependent at Week 24.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Momelotinib (MMB) | Ruxolitinib (RUX)
Number analyzed (Participants) | 215 | 217
Participants
  Dependent | 65 | 87
  Nondependent | 150 | 130
Statistical Analysis 1: Comparison: Momelotinib (MMB) vs Ruxolitinib (RUX); Test type: Superiority; p = 0.019, Cochran-Mantel-Haenszel; Proportion Difference - Stratified CMH = -0.10, 95% CI 2-sided [-0.19 to -0.02] — A smaller proportion represents larger benefit

ADVERSE EVENTS:
Time Frame: Serious and other Adverse events were recorded that occurred from initiation of investigational product (IP) until 30 days after the last administration of IP regardless of cause or relationship. Serious events are monitored up to 12 weeks and all-cause mortality was assessed for up to 5 years.
Description: The safety population did not include 2 patients (one on MMB and one on RUX) who were not dosed, hence affecting the total number of patients at risk.
Arm/Group | Momelotinib (MMB) | Ruxolitinib (RUX) | MMB to MMB | RUX to MMB
All-Cause Mortality (participants affected / at risk) | 8/214 | 6/216 | 44/171 | 54/197
Serious Adverse Events (participants affected / at risk) | 49/214 | 39/216 | 79/171 | 79/197
Other Adverse Events (participants affected / at risk) | 197/214 | 206/216 | 153/171 | 188/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Momelotinib (MMB) (N=214) | Ruxolitinib (RUX) (N=216) | MMB to MMB (N=171) | RUX to MMB (N=197)
Anaemia (Blood and lymphatic system disorders) | 4 | 8 | 7 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Splenic haematoma (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 3 | 0
Splenic thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 4
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 1 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 1 | 3 | 4
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2 | 1
Cardiac failure (Cardiac disorders) | 2 | 0 | 5 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 2 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Cataract nuclear (Eye disorders) | 0 | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0 | 4
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Visceral venous thrombosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 2
Death (General disorders) | 1 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 1
Mucosal haemorrhage (General disorders) | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 3 | 3 | 1
Sudden death (General disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Abdominal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 2 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 2
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 2
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 3 | 0
Neuroborreliosis (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 3 | 16 | 9
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 2 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 2 | 1 | 6 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Serratia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Tetanus (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 5
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Langerhans cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Mantle cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Ovarian clear cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Primary myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Cerebellar stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral venous thrombosis (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 3 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1
Coma (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 3 | 4
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 3 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 3
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Breast hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 3 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Momelotinib (MMB) (N=214) | Ruxolitinib (RUX) (N=216) | MMB to MMB (N=171) | RUX to MMB (N=197)
Abdominal pain (Gastrointestinal disorders) | 21 | 24 | 13 | 26
Alanine aminotransferase increased (Investigations) | 10 | 10 | 5 | 11
Anaemia (Blood and lymphatic system disorders) | 30 | 79 | 38 | 29
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 10 | 10 | 13
Asthenia (General disorders) | 12 | 16 | 13 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 10 | 10 | 19
Blood creatinine increased (Investigations) | 9 | 2 | 10 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 15 | 4 | 12
Constipation (Gastrointestinal disorders) | 21 | 15 | 13 | 18
Contusion (Injury, poisoning and procedural complications) | 16 | 10 | 9 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 17 | 23 | 34
Decreased appetite (Metabolism and nutrition disorders) | 11 | 13 | 15 | 15
Diarrhoea (Gastrointestinal disorders) | 36 | 42 | 30 | 37
Dizziness (Nervous system disorders) | 34 | 25 | 17 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 17 | 14 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 14 | 8 | 12
Fatigue (General disorders) | 31 | 26 | 17 | 38
Flushing (Vascular disorders) | 13 | 1 | 1 | 3
Headache (Nervous system disorders) | 38 | 43 | 13 | 24
Hypertension (Vascular disorders) | 9 | 19 | 10 | 18
Hyperuricaemia (Metabolism and nutrition disorders) | 10 | 7 | 11 | 14
Hypotension (Vascular disorders) | 18 | 1 | 6 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 11 | 1 | 5
Nasopharyngitis (Infections and infestations) | 9 | 16 | 7 | 14
Nausea (Gastrointestinal disorders) | 33 | 8 | 16 | 39
Neutropenia (Blood and lymphatic system disorders) | 9 | 14 | 7 | 7
Oedema peripheral (General disorders) | 10 | 13 | 16 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 18 | 11 | 19
Paraesthesia (Nervous system disorders) | 15 | 7 | 6 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 20 | 12 | 15 | 28
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 11 | 12 | 20
Pyrexia (General disorders) | 12 | 14 | 15 | 14
Rash (Skin and subcutaneous tissue disorders) | 9 | 5 | 10 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 40 | 62 | 29 | 39
Upper respiratory tract infection (Infections and infestations) | 12 | 14 | 18 | 18
Urinary tract infection (Infections and infestations) | 10 | 9 | 19 | 19
Vomiting (Gastrointestinal disorders) | 20 | 7 | 8 | 11
Night sweats (Skin and subcutaneous tissue disorders) | 8 | 9 | 12 | 17
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 7 | 12 | 8 | 11
Fall (Injury, poisoning and procedural complications) | 6 | 4 | 9 | 8
Bronchitis (Infections and infestations) | 4 | 5 | 8 | 11
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 3 | 4 | 11
Insomnia (Psychiatric disorders) | 4 | 6 | 11 | 6
Aspartate aminotransferase increased (Investigations) | 7 | 5 | 3 | 10
Pneumonia (Infections and infestations) | 1 | 4 | 4 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 4 | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements varied with individual investigators, but did not prohibit any investigator from publishing. Investigators were not to publish results of the study until a period of time (eg. 2 years) following completion of the trial at all participating institutions but could do so earlier with consent of the Sponsor.